CLINICAL TRIAL: NCT02145351
Title: Rate-Adaptive Atrial Pacing In Diastolic Heart Failure (RAPID-HF)
Brief Title: Efficacy Study of Pacemakers to Treat Slow Heart Rate in Patients With Heart Failure
Acronym: RAPID-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Barry Borlaug, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13-008306
Record Dates: First submitted 2014-05-20; First posted 2014-05-22 (Estimated); Results first posted 2023-04-05 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-03

CONDITIONS: Heart Failure With a Preserved Ejection Fraction; Heart Failure, Diastolic; Chronotropic Incompetence
Keywords: HFpEF; Heart failure; Heart failure with preserved ejection fraction; Chronotropic incompetence
MeSH Terms: conditions — Heart Failure, Diastolic; Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Pacing off first, then pacing on (Active Comparator): No-pacing on for the first for 4 weeks, followed by 4 week washout period, and then cross-over to pacing on for an additional 4 weeks.
  Interventions: Device: Rate adaptive atrial pacing using a dual-chamber pacemaker; Device: Pacemaker system will be implanted but set to Pacing Off.
- Pacing on first, then pacing off (Experimental): Pacing on for the first for 4 weeks, followed by 4 week washout period, and then cross-over to pacing off for an additional 4 weeks
  Interventions: Device: Rate adaptive atrial pacing using a dual-chamber pacemaker; Device: Pacemaker system will be implanted but set to Pacing Off.

INTERVENTIONS:
Device: Rate adaptive atrial pacing using a dual-chamber pacemaker — The Azure XT DR is a permanent, dual-chamber cardiac pacemaker with the ability to continuously monitor and record patient activity, and respond to activity by pacing faster and increasing the heart rate (rate adaptive atrial pacing). It will be programmed in AAIR mode to pace the right atrium. The leads will be placed in the right atrium and right ventricle using CapSureFix model 5086.
  Other Names: Medtronic Azure XT DR MRI pacemaker model W1DR01; Medtronic CapSureFix MRI model 5086
Device: Pacemaker system will be implanted but set to Pacing Off. — The identical pacing system will be implanted, but will be set to Pacing Off.
  Other Names: Medtronic Azure XT DR MRI model W1DR01; Medtronic CapSureFix MRI model 5086

SUMMARY:
Determine the impact of restoring normal heart rate response during exercise and daily activity in patients with heart failure and a preserved ejection fraction (HFpEF) and chronotropic incompetence (CI).

ELIGIBILITY:
Inclusion Criteria

1. Age >18 years and able to provide informed consent to enroll in the trial, or consent through a legal guardian or power of attorney.
2. Previous clinical diagnosis of HF with current NYHA Class II-III symptoms
3. At least one of the following: Hospitalization for decompensated HF, Acute treatment for HF with intravenous loop diuretic or hemofiltration, Chronic treatment with a loop diuretic for control of HF symptoms + left atrial enlargement on echocardiography or E/e' ratio (≥14 average, ≥15 septal ) on echocardiography, Resting PCWP >15 mm Hg or LV end-diastolic pressure >18 mmHg at catheterization for dyspnea and/or exercise PCWP/LV end-diastolic pressure >25 mmHg, or Elevated NT-proBNP level (≥300 pg/ml )
4. Left ventricular EF ≥40% within 12 months with clinical stability
5. Stable cardiac medical therapy for ≥30 days
6. Sinus rhythm
7. Chronotropic incompetence on recent (within 6 months) clinical or screening exercise test, defined as heart rate reserve (HRR) <0.80 or <0.62 if on beta blockers
8. Meet both screening criteria on clinically-performed cardiopulmonary exercise testing within 12 months.

Exclusion Criteria

1. Inability to exercise, or non-cardiac condition that precludes exercise testing
2. Any contraindication to a pacemaker system
3. Non-cardiac condition limiting life expectancy to less than one year
4. Significant left sided structural valve disease (>mild stenosis, >moderate regurgitation)
5. Hypertrophic cardiomyopathy
6. Infiltrative or inflammatory myocardial disease (amyloid, sarcoid)
7. Pericardial disease
8. Non-group 2 pulmonary arterial hypertension
9. Chronic stable exertional angina
10. Acute coronary syndrome or revascularization within 60 days
11. Other clinically important causes of dyspnea
12. Atrial fibrillation
13. PR interval >210 msec
14. Resting heart rate (HR) > 100 bpm
15. A history of reduced ejection fraction (EF<40%)
16. Advanced chronic kidney disease (GFR < 20 ml/min/1.73m2 by modified MDRD equation)
17. Women of child bearing potential without negative pregnancy test and effective contraception
18. Severe anemia (Hemoglobin <10 g/dL)
19. Severe hepatic disease
20. Complex congenital heart disease
21. Listed for cardiac transplantation
22. Other class I indications for pacing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-04-07 (Actual); Primary Completion 2022-05-09 (Actual); Study Completion 2022-05-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barry Borlaug, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reddy YNV, Koepp KE, Carter R, Win S, Jain CC, Olson TP, Johnson BD, Rea R, Redfield MM, Borlaug BA. Rate-Adaptive Atrial Pacing for Heart Failure With Preserved Ejection Fraction: The RAPID-HF Randomized Clinical Trial. JAMA. 2023 Mar 14;329(10):801-809. doi: 10.1001/jama.2023.0675. PMID 36871285
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Three subjects did not return for baseline testing following pacemaker implantation, leaving a total of 29 patients who were randomized into the study.
Groups:
- Pacing Off First, Then Pacing on: Subjects who received pacing off in either the first or last 4 weeks of the study
  Pacing off for the first for 4 weeks, followed by 4 week washout period, and then cross-over to pacing on for an additional 4 weeks.
  Rate adaptive atrial pacing using a dual-chamber pacemaker: The Azure XT DR is a permanent, dual-chamber cardiac pacemaker with the ability to continuously monitor and record patient activity, and respond to activity by pacing faster and increasing the heart rate (rate adaptive atrial pacing). It will be programmed in AAIR mode to pace the right atrium. The leads will be placed in the right atrium and right ventricle using CapSureFix model 5086.
  Pacemaker system implanted but set to Pacing Off.: The identical pacing system will be implanted, but will be set to Pacing Off.
- Pacing on First, Then Pacing Off: Subjects who received pacing on either the first or last 4 weeks of the study
  Pacing on for the first for 4 weeks, followed by 4 week washout period, and then cross-over to pacing off for an additional 4 weeks
  Rate adaptive atrial pacing using a dual-chamber pacemaker: The Azure XT DR is a permanent, dual-chamber cardiac pacemaker with the ability to continuously monitor and record patient activity, and respond to activity by pacing faster and increasing the heart rate (rate adaptive atrial pacing). It will be programmed in AAIR mode to pace the right atrium. The leads will be placed in the right atrium and right ventricle using CapSureFix model 5086.
  Pacemaker system implanted but set to Pacing Off.: The identical pacing system will be implanted, but will be set to Pacing Off.
- Pacemaker Implantation: All subjects who had a pacemaker implanted 4 weeks prior to randomization
Period: Pacemaker Implantation (4 Weeks)
Arm/Group | Pacing Off First, Then Pacing on | Pacing on First, Then Pacing Off | Pacemaker Implantation
Started | 0 | 0 | 32
Completed | 0 | 0 | 32
Not Completed | 0 | 0 | 0
Period: First Intervention (4 Weeks)
Arm/Group | Pacing Off First, Then Pacing on | Pacing on First, Then Pacing Off | Pacemaker Implantation
Started | 15 | 14 | 0
Completed | 15 | 14 | 0
Not Completed | 0 | 0 | 0
Period: Washout (4 Weeks)
Arm/Group | Pacing Off First, Then Pacing on | Pacing on First, Then Pacing Off | Pacemaker Implantation
Started | 15 | 14 | 0
Completed | 15 | 14 | 0
Not Completed | 0 | 0 | 0
Period: Second Intervention (4 Weeks)
Arm/Group | Pacing Off First, Then Pacing on | Pacing on First, Then Pacing Off | Pacemaker Implantation
Started | 15 | 14 | 0
Completed | 15 | 14 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pacing Off First, Then Pacing on | Pacing on First, Then Pacing Off | Total
Number analyzed (Participants) | 15 | 14 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.5 (12.2) | 65.4 (6.4) | 66.0 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 7 | 9 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 15 | 14 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 14 | 29

OUTCOME MEASURES:

1. Primary Outcome: Change in Oxygen Consumption (VO2) at Ventilatory Anaerobic Threshold (VAT)
Description: Maximal effort cardiopulmonary exercise testing was performed on a treadmill after 4 weeks of pacing-on and after 4 weeks of pacing-off to measure volumes of oxygen consumed (VO2). Change in VO2 at anaerobic threshold (VO2,AT) determined by the V-Slope method as the point of disproportionate rise in VCO2 relative to VO2 as measured in ml/kg/min.
Time Frame: baseline, after 4 weeks of treatment
Measure: Mean (Standard Deviation); unit: ml/kg/min
Groups:
- Pacing Off: Subjects who received pacing off in either the first or last 4 weeks of the study
- Pacing on: Subjects who received pacing on either the first or last 4 weeks of the study
Arm/Group | Pacing Off | Pacing on
Number analyzed (Participants) | 29 | 29
ml/kg/min | 10.4 (2.9) | 10.7 (2.6)

2. Secondary Outcome: Peak Aerobic Capacity (Peak VO2)
Description: Determined as the mean of values obtained over the final 30 seconds of exercise. Maximal effort cardiopulmonary exercise testing was performed on a treadmill after 4 weeks of pacing-on and after 4 weeks of pacing-off to measure volumes of oxygen consumed (VO2). As measured in ml/kg/min.
Time Frame: 4 weeks after pacemaker activation
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | Pacing Off | Pacing on
Number analyzed (Participants) | 29 | 29
ml/kg/min | 16.5 (4.3) | 16.8 (4.1)

3. Secondary Outcome: Ventilatory Efficiency (VE/VCO2)
Description: Determined as the nadir of VE/VCO2 ratio during exercise. Maximal effort cardiopulmonary exercise testing was performed on a treadmill after 4 weeks of pacing-on and after 4 weeks of pacing-off to measure volumes of oxygen consumed (VO2).
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Pacing Off | Pacing on
Number analyzed (Participants) | 29 | 29
ratio | 34.2 (6.6) | 34.9 (6.3)

4. Secondary Outcome: Change in Plasma N-terminal Pro B-type Natriuretic Peptide (NT-proBNP)
Description: Change in plasma NT-proBNP as measured in pg/mL. Natriuretic peptides are substances made by the heart. A main type of these substances is NT-proBNP. Elevated levels can mean the heart isn't pumping as much blood the body needs.
Time Frame: baseline, after 4 weeks of treatment
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Pacing Off | Pacing on
Number analyzed (Participants) | 29 | 29
pg/mL | -88.0 (390) | -36.0 (255)

5. Secondary Outcome: Change in Kansas City Cardiomyopathy Questionnaire (KCCQ) Overall Summary Score
Description: Change from baseline in KCCQ-overall summary score was reported. KCCQ was a 23-item, self-administered questionnaire that measure the participant's perception of their health status, including their heart failure (HF) symptoms, impact on physical and social function and how their HF impacts the quality of life. KCCQ quantifies 7 domains: physical limitations (6 items), symptom stability (1 item), symptom frequency (4 items), symptom burden (3 items), self-efficacy (2 items), quality of life (3 items) and social limitations (4 items). Scores were generated for each domain and scaled from 0 to 100, with 0 denoting the worst and 100 the best possible status. KCCQ- overall summary score was average of domains- physical limitation, total symptoms (average of symptom frequency and symptom burden), quality of life, and social limitation, and transformed to a single score which ranged from 0 (worst) -100 (the best possible status), where the higher score reflected better health status.
Time Frame: baseline, after 4 weeks of treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pacing Off | Pacing on
Number analyzed (Participants) | 29 | 29
score on a scale | 4.7 (16.4) | 3.8 (20.2)

6. Other Pre Specified Outcome: Mean Peak Heart Rate (HR)
Description: Determined as the maximum heart rate . Heart rate (or pulse rate) is the frequency of the heartbeat measured by the number of contractions of the heart per minute (beats per minute, or bpm).
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Pacing Off | Pacing on
Number analyzed (Participants) | 29 | 29
bpm | 109 (21) | 123 (15)

ADVERSE EVENTS:
Time Frame: Adverse Events were assessed for all subjects during Pacemaker implantation (4 weeks), first treatment period (4 weeks), washout period (4 weeks), and second treatment period (4 weeks) for a total of approximately 16 weeks.
Groups:
- Pacing Off: Subjects who received pacing off in either the first or last 4 weeks of the study
  Pacemaker system implanted but set to Pacing Off.: The identical pacing system will be implanted, but will be set to Pacing Off.
- Pacing on: Subjects who received pacing on either the first or last 4 weeks of the study
  Rate adaptive atrial pacing using a dual-chamber pacemaker: The Azure XT DR is a permanent, dual-chamber cardiac pacemaker with the ability to continuously monitor and record patient activity, and respond to activity by pacing faster and increasing the heart rate (rate adaptive atrial pacing). It will be programmed in AAIR mode to pace the right atrium. The leads will be placed in the right atrium and right ventricle using CapSureFix model 5086.
- Pacemaker Implantation: Subjects who experience adverse events during pacemaker implantation procedure only. This would be the timeframe after consent and prior to randomization to either pacing off or pacing on.
- Washout Period: After first intervention, both pacing off and pacing on groups will have a 4 week washout period when the pacemaker is turned off.
Arm/Group | Pacing Off | Pacing on | Pacemaker Implantation | Washout Period
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/29 | 0/32 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/29 | 1/32 | 0/29
Other Adverse Events (participants affected / at risk) | 8/29 | 7/29 | 5/32 | 0/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pacing Off (N=29) | Pacing on (N=29) | Pacemaker Implantation (N=32) | Washout Period (N=29)
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pacing Off (N=29) | Pacing on (N=29) | Pacemaker Implantation (N=32) | Washout Period (N=29)
Chest discomfort/palpitations (Cardiac disorders) | 1 | 5 | 0 | 0
Pacing lead induced tricuspid regurgitation (Cardiac disorders) | 0 | 0 | 1 | 0
Upper extremity deep venous thrombosis (Cardiac disorders) | 0 | 0 | 1 | 0
Incision site reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 0
Dizziness (Nervous system disorders) | 3 | 0 | 0 | 0
Worsening fatigue (General disorders) | 2 | 1 | 0 | 0
Non pacemaker infection (Infections and infestations) | 2 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-30): https://cdn.clinicaltrials.gov/large-docs/51/NCT02145351/Prot_SAP_000.pdf